CLINICAL TRIAL: NCT07407972
Title: Effect of Optıc Nerve Dıameter ın Tymphanoplasty Surgery Performed ın Lateral Head Posıtıon Under General Anesthesia
Brief Title: Effect of Optıc Nerve Dıameter ın Tymphanoplasty Surgery Performed ın Lateral Head Posıtıon
Acronym: ONSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, sermın emınoglu, associate professor, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-KAEK-25 2020/01-12
Record Dates: First submitted 2026-01-29; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Optic Nerve Diameter; Intracranial Pressure Increase
Keywords: tympanoplasty; lateral position; optic nerve diameter; intracranial pressure; headache and sore throat
MeSH Terms: conditions — Intracranial Hypertension; Headache; Pharyngitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ONSD Measurement (Other): ONSD measurements were taken in three time intervals by the anesthesiologist: transverse and sagittal planes. Both ONSDs were recorded by ultrasound at T1: 5 min in supine position, T2: end of the procedure with head in lateral position, and T3: supine position before extubation.
  Interventions: Diagnostic Test: optic nerve diameter

INTERVENTIONS:
Diagnostic Test: optic nerve diameter — optic nerve diameter measurement

SUMMARY:
Studies exist to determine the effect of laparoscopic surgical procedures on increased intra-abdominal pressure; these studies include optic nerve sheath diameter (ONSD) measurement in various positions such as trendelenburg and prone, and the effect of the laryngoscope used in intubation on increased intracranial pressure. In these situations, changes in cerebral blood flow and intracranial pressure may occur due to impaired neck venous return. There are no studies in the literature regarding increased osd and consequently increased intracranial pressure in lateral head position.ultrasound for ONSD measurement is a non-invasive, rapid, and easily applicable method for diagnosing changes in intracranial pressure. In tympanoplasty surgeries, the head and neck remain in a lateral position, and venous return in the surgical field may sometimes be compressed due to the procedure. The aim of this study is to determine the effect of lateral head position and variables such as demographic data and surgical duration on increased intracranial pressure. Methods: Patients over 18 years of age, classified as asa ı and ıı, undergoing tympanoplasty surgery under general anesthesia in the lateral head and neck position will be included in the study. Patients' vital signs (arterial blood pressure, heart rate, spo2, and etco2) will be monitored regularly in the operating room before and after surgery. Demographic data (age, gender, weight, height), surgery duration, and postoperative complications will also be recorded. Anesthesia will be administered with 2-4 mg/kg propofol, 0.6 mg/kg rocuronium, and 1-2 mcg/kg fentanyl for induction, and sevoflurane for maintenance. Following intubation, onstitial lateral head and neck (onsd) measurements will be taken by the anesthesiologist at three time intervals (in transverse and sagittal planes). Both onsds will be recorded by ultrasound: T1: 5 minutes in the supine position, T2: at the end of the procedure with the head in the lateral position, and T3: before extubation in the supine position. Postoperative headache and neck pain will be inquired about after waking up and at 1., 6., and 24. hours later.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age Patients undergoing tympanoplasty surgery under general anesthesia Patients with ASA I or II Patients scheduled for surgery in the lateral head and neck position

Exclusion Criteria:

* Patients who will have neck dissection,
* Patients who have undergone other procedures that may cause changes in -intracranial pressure,
* Patients under 18 years of age,
* Patients who cannot communicate,
* Patients with glaucoma and eye disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
The effect of lateral head position on intracranial pressure | 2 years
  The effect of lateral head positioning on intracranial pressure will be determined by measuring the diameter of the optic nerve sheath under ultrasound guidance.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa yüksek ihtisas eğitim ve araştırma hastanesi BURSA, Bursa, Türkiye, Bursa, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and results can be shared.
Supporting Information: Study Protocol

REFERENCES:
- [Result] Altiparmak B, Pinarbasi A, Korkmaz Toker M, Uysal AI, Turan M. Neck extension during thyroidectomy: effects on early postoperative cognitive function and optic nerve sheath diameter- a randomized controlled trial. BMC Anesthesiol. 2025 Dec 1;26(1):15. doi: 10.1186/s12871-025-03507-y. PMID 41327017

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT07407972/Prot_SAP_000.pdf